CLINICAL TRIAL: NCT05543161
Title: "Peripheral Blood Dipeptidylpeptidase IV (CD26) Positive Leukemic Stem Cells in Chronic Myeloid Leukemia as a Diagnostic Marker"
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Rowaida Moahmed Mohamed, Clinical pathology specialist , Sohag general hospital, Sohag University
Other Study IDs: Soh-Med-22-09-10
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Chronic Myeloid Leukemia, Chronic Phase
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood sample for immunophenotyping
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic myeloid leukemia (CML) is a stem cell (SC) neoplasm which originates from an incomplete process of differentiation of the hematopoietic stem cells (HSCs) to the adult cells which lead to accumulation of their immature form into the BM and the peripheral blood. It is characterized by the reciprocal translocation. The resulting oncoprotein, BCR/ABL1, is considered essential for the initiation and manifestation of the disease . In CML, leukemic stem cell (LSC) supposedly resides within the CD45+/ CD34+/CD38-/Lin- fraction of the leukemic clone (3). However, normal hematopoietic SC also exhibit this phenotype so that additional markers are required to discriminate CML LSC from normal SC. CD34+/CD38-/Lin- CML LSC specifically co-express dipeptidylpeptidase IV(DPPIV=CD26). This enzyme disrupts LSC-niche interactions by degrading stroma derived factor-1 (SDF-1). Moreover, CD26 is a robust biomarker for the quantification and isolation of CML LSC (4). It was reported that CD26+ LSCs were significantly correlated with BCR-ABL1 transcript level at diagnosis and after three months of treatment with tyrosine kinase inhibitor (TKI) .

ELIGIBILITY:
Inclusion Criteria:

* : All suspected patients for CML diagnosis aged more than 18 years who presented with high white blood cells(WBCs) count , marked shift to left in peripheral blood with or without splenomegaly .

Exclusion Criteria:

* Patients on treatment or presence of blasts in peripheral blood sample.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All suspected patients for CML diagnosis aged more than 18 years who presented with high white blood cells(WBCs) count , marked shift to left in peripheral blood with or without splenomegaly .
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Peripheral Blood Dipeptidylpeptidase IV (CD26) | 1 year
  to detect CD26+ LSCs by flow cytometry for accurate diagnosis of CML patients from peripheral blood sample to reduce the need for Bone Marrow aspiration.

CONTACTS AND LOCATIONS:
Overall Officials: Eid, Principal Investigator — Sohag univerisity
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] Lane SW, Scadden DT, Gilliland DG. The leukemic stem cell niche: current concepts and therapeutic opportunities. Blood. 2009 Aug 6;114(6):1150-7. doi: 10.1182/blood-2009-01-202606. Epub 2009 Apr 28. PMID 19401558
- [Background] Ebian HF, Abdelnabi AM, Abdelazem AS, Khamis T, Fawzy HM, Hussein S. Peripheral blood CD26 positive leukemic stem cells as a possible diagnostic and prognostic marker in chronic myeloid leukemia. Leuk Res Rep. 2022 May 9;17:100321. doi: 10.1016/j.lrr.2022.100321. eCollection 2022. PMID 35602932
- [Background] Waumans Y, Baerts L, Kehoe K, Lambeir AM, De Meester I. The Dipeptidyl Peptidase Family, Prolyl Oligopeptidase, and Prolyl Carboxypeptidase in the Immune System and Inflammatory Disease, Including Atherosclerosis. Front Immunol. 2015 Aug 7;6:387. doi: 10.3389/fimmu.2015.00387. eCollection 2015. PMID 26300881
- [Background] Lee SA, Kim YR, Yang EJ, Kwon EJ, Kim SH, Kang SH, Park DB, Oh BC, Kim J, Heo ST, Koh G, Lee DH. CD26/DPP4 levels in peripheral blood and T cells in patients with type 2 diabetes mellitus. J Clin Endocrinol Metab. 2013 Jun;98(6):2553-61. doi: 10.1210/jc.2012-4288. Epub 2013 Mar 28. PMID 23539735